CLINICAL TRIAL: NCT04079855
Title: Diet-induced Modification of Sweet Taste Perception and Preference
Brief Title: Monell USDA Taste Test Study
Acronym: MUTT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Baer (U.S. Federal Agency)
Collaborators: Monell Chemical Senses Center (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, David Baer, Supervisory Reserach Physiologist, USDA Beltsville Human Nutrition Research Center
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HS65 - MUTT Study; 5U01DC013529 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention is of foods which will look identical. Volunteers will know the color of their treatment assignment but not the actual identity of their treatment. The investigators will use a double masking protocol in which investigators and outcome assessors (study staff who collect primary and secondary measures and data analysts) will not know the treatment assignments or treatment coding (color coded) scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diet composition 1 (Experimental): A diet with a specified macronutrient composition different from arms 2 and 3.
  Interventions: Other: Diet composition 1
- Diet composition 2 (Experimental): A diet with a specified macronutrient composition different from arms 1 and 3.
  Interventions: Other: Diet composition 2
- Diet composition 3 (Experimental): A diet with a specified macronutrient composition different from arms 1 and 2, based on the current information about the US macronutrient composition.
  Interventions: Other: Diet composition 3

INTERVENTIONS:
Other: Diet composition 1 — A diet with a specified macronutrient composition different from arms 2 and 3.
  Arms: Diet composition 1
Other: Diet composition 2 — A diet with a specified macronutrient composition different from arms 1 and 3.
  Arms: Diet composition 2
Other: Diet composition 3 — A diet with a specified macronutrient composition different from arms 1 and 2, based on the current information about the US macronutrient composition.
  Arms: Diet composition 3

SUMMARY:
Overconsumption of carbohydrates has been implicated as a cause of significant public health problems including obesity and diabetes. The most effective approach to alter dietary pattern and improve public health is unknown. Gradual and abrupt changes in dietary pattern have been tried in small, uncontrolled trials, but it is not clear which approach is most effective. The primary objective of this study is to evaluate different approaches to changing dietary pattern for altering flavor perception in foods and beverages and for altering preference for flavor.

DETAILED DESCRIPTION:
This comprehensive, well-controlled diet study aims to evaluate and compare different approaches to alter dietary pattern, especially macronutrient profile. The investigators propose a prospective, randomized trial that is designed to overcome the above limitations to test the hypothesis that changing dietary macronutrient profile can change taste perception and food preference. Data from this study will provide information that policy makers, regulators, and the food industry can use to develop successful approaches (gradual or otherwise) for providing healthy diets in the marketplace.

ELIGIBILITY:
Exclusion criteria Younger than 25 years old and older than 80 years old at the beginning of the intervention.

Have body weight less than 110 lbs.

Known (self-reported) allergy or adverse reaction to study foods or ingredients

Added sugars intake at baseline < 10% of total energy.

A dietary pattern inconsistent with the dietary intervention (i.e., vegan, vegetarian, extremes of protein, fat, carbohydrate intake).

Body mass index less than 18 or greater than 40 kg/m2

Women who have given birth during the previous 12 months, are pregnant, are lactating, or plan to become pregnant during the study.

Use of appetite suppressants or other anti-obesity medication during the past 6 months.

History of bariatric or certain other surgeries related to weight control.

History or presence of diabetes, kidney disease, liver disease, certain cancers, gout, hyperthyroidism, untreated or unstable hypothyroidism, gastrointestinal disease, pancreatic disease, other metabolic diseases, malabsorption syndromes, phenylketonuria, or endocrine disorders that may interfere with the study outcomes.

Individuals with any gastrointestinal issues, including bariatric surgery, inflammatory bowel disease, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, nutrient malabsorption disease, or Crohn's Disease Smokers or other tobacco/marijuana users (within 6 months prior to the study).

History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians).

Known taste or smell disorders, including weak or absent sense of taste or smell (screening procedures include a basic taste and smell sensitivity tests), abnormal taste in the mouth (e.g., bitter or metallic "phantom" tastes), or other taste abnormality.

Use of medications within one month prior to the study that moderately to severely affect taste.

Tested positive for COVID-19 in the past 4 weeks.

Volunteers who have lost or gained >10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 12 months.

Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion); evaluated using USAUDIT.

Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Unable or unwilling to give informed consent or communicate with study staff.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Taste intensity of food | Month 1
  Rating taste intensity from barely detectable to strong using a general labeled magnitude scale. The name of the scale is the general labeled magnitude scale. The value of the response is recorded on the scale as "barely detectable", "weak", "moderate, strong", "very strong", and "strongest imaginable sensation of any kind." None of these responses is considered better or worse than any other.
Taste intensity of food | Month 2
  Rating taste intensity from barely detectable to strong using a general labeled magnitude scale. The name of the scale is the general labeled magnitude scale. The value of the response is recorded on the scale as "barely detectable", "weak", "moderate, strong", "very strong", and "strongest imaginable sensation of any kind." None of these responses is considered better or worse than any other.
Taste intensity of food | Month 3
  Rating taste intensity from barely detectable to strong using a general labeled magnitude scale. The name of the scale is the general labeled magnitude scale. The value of the response is recorded on the scale as "barely detectable", "weak", "moderate, strong", "very strong", and "strongest imaginable sensation of any kind." None of these responses is considered better or worse than any other.
Taste intensity of food | Month 4
  Rating taste intensity from barely detectable to strong using a general labeled magnitude scale. The name of the scale is the general labeled magnitude scale. The value of the response is recorded on the scale as "barely detectable", "weak", "moderate, strong", "very strong", and "strongest imaginable sensation of any kind." None of these responses is considered better or worse than any other.
Taste intensity of food | Month 6
  Rating taste intensity from barely detectable to strong using a general labeled magnitude scale. The name of the scale is the general labeled magnitude scale. The value of the response is recorded on the scale as "barely detectable", "weak", "moderate, strong", "very strong", and "strongest imaginable sensation of any kind." None of these responses is considered better or worse than any other.
Taste preference | Month 1
  Most liked concentration. Foods will be scaled as g flavor/100 g food.
Taste preference | Month 2
  Most liked concentration. Foods will be scaled as g flavor/100 g food.
Taste preference | Month 3
  Most liked concentration. Foods will be scaled as g flavor/100 g food.
Taste preference | Month 4
  Most liked concentration. Foods will be scaled as g flavor/100 g food.
Taste preference | Month 6
  Most liked concentration. Foods will be scaled as g flavor/100 g food.

SECONDARY OUTCOMES:
Diet-related adverse events | Daily during the Baseline (Month 1), Months 2-6
  Adverse events related to the diet tabulated by study-arm and severity.
Diet-related early discontinuation from intervention | Daily during the Baseline (Month 1), Months 2-6
  Subject withdraws citing issues with the study diet, or investigators withdraw the subject from the study due to concerns over how the subject reacts to the study diet.

OTHER OUTCOMES:
Glucose | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  Glucose is a sugar that circulates in the blood and is used as an energy source for many cells. Glucose will be measured to determine how the treatment is affecting blood glucose regulation. Glucose is measured in units of mg/dL.
Insulin | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  Insulin is a hormone that helps control blood glucose concentration. Insulin will be measured to determine how the treatment is affecting blood glucose regulation. Insulin is measured in units of microIU/mL.
c-peptide | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  c-peptide is a peptide that is formed during the production of insulin. C-peptide will be measured to determine how the treatment is affecting insulin response and blood glucose regulation. c-peptide is measured in units of ng/mL.
Glucagon | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  Glucagon is a hormone that helps control blood glucose concentration. Glucagon will be measured to determine how the treatment is affecting blood glucose regulation. Glucagon is measured in units of pg/mL.
Glucagon-like peptide-1 (GLP-1) | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  GLP-1 is a hormone that helps control blood glucose concentration. GLP-1 will be measured to determine how the treatment is affecting blood glucose regulation. GLP-1 is measured in units of pg/mL.
Anandamide | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  Anandamide is the precursor of a class of physiologically active substances which are involved in brain chemistry. Anandamide will be measured to determine how the treatment is affecting blood compounds that are associated with reward. Anandamide is measured in units of ng/mL.
2-arachidonyl glycerol (2-AG) | Baseline (Month 1) week 3 or 4, Months 2-4, Month 6
  2-AG is the precursor of a class of physiologically active substances which are involved in brain chemistry. 2-AG will be measured to determine how the treatment is affecting blood compounds that are associated with reward. 2-AG is measured in units of ng/mL.
Sweet taste receptors genotype | Baseline month (once)
  Genotyping describes the genetic make-up. The known variants of sweet receptor subunit TAS1R3 will be genotyped. Genotype will be measured as a specific sequence of the nucleobases cytosine, guanine, adenine and thymine.
Body weight | Baseline, Months 2-4 M-F, Month 6 at end of study
  Body weight is the mass of a person. Body weight is measured wearing street clothes without shoes or other heavy items in the pockets. Body weight is used to adjust energy intake to maintain weight maintenance. Body weight is measured in kg.
Waist circumference | Screening and Month 6 at end of study
  Waist circumference is the distance around an individual at a specific location. Waist circumference is measured in cm.
Blood pressure | Screening and Month 6 at end of study
  Blood pressure is a measure of the pressure produced by the heart on the walls of the blood vessels at different times during the heartbeat. Blood pressure is measured in mm Hg (mercury).
Power of Food Scale | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior. There are 15 items on the questionnaire. Each item is recorded as a 5-point Likert scale with a value of 1, 2, 3, 4, or 5 corresponding to "I don't agree", "I agree a little", "I agree somewhat", "I agree quite a bit, and "I strongly agree". A total score is determined as the sum of the responses. None of these responses is considered better or worse than any other.
Emotional Eating Scale | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior. There are 25 items on the questionnaire. Each item is recorded as a 5-point Likert scale with a value of 1, 2, 3, 4, or 5 corresponding to "no desire to eat", "a small desire to eat", "a moderate desire to eat", "a strong urge to eat", or "an overwhelming urge to eat." A total score is determined as the sum of the responses. None of these responses is considered better or worse than any other.
Three Factor Eating Questionnaire | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior.
Dutch Eating Behaviour Questionnaire | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior.
Yale Food Addiction Scale | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior. There are 16 items on the questionnaire that are scored as a 5-point Likert scale with a value of 0, 1, 2, 3, or 4, corresponding to "never", "once a month", "2-4 times a month", "2-3 times a week", or "4 or more times or daily." There is 1 item on the questionnaire that is scored as a 5-point Likert scale with a value of 0, 1, 2, 3, or 4, corresponding to "1 or fewer times", "2 times", "3 times", "4 times", or "5 or more times." There are 8 items scored as "no" (0) or "yes" (1). A total score is determined as the sum of the responses. None of these responses is considered better or worse than any other.
Barrat Impulsiveness Scale | Baseline and Month 6 end of study
  A questionnaire that measures factors related to food preference and eating behavior. There are 11 items on the questionnaire that are scored as a 4-point Likert scale with a value of 1, 2, 3, or 4 corresponding to "rarely/never", "occasionally", "often", or "almost always/always." A total score is determined as the sum of the responses. None of these responses is considered better or worse than any other.
Dietary Satisfaction Questionnaire | Baseline, weekly during Months 3-5, and Month 6 end of intervention
  A questionnaire that measures factors related to food preference and eating behavior.
Food Craving Inventory | Baseline, weekly during Months 3-5, and Month 6 end of intervention
  A questionnaire that measures factors related to food preference and eating behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wise, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States